CLINICAL TRIAL: NCT00045747
Title: Phase II Study of UCN-01 in Combination With Fluorouracil in Advanced Pancreatic Cancer
Brief Title: UCN-01 and Fluorouracil in Treating Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000257125; MSKCC-02049; NCI-5509
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2004-08

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; recurrent pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 7-hydroxystaurosporine; Fluorouracil

INTERVENTIONS:
Drug: 7-hydroxystaurosporine
Drug: fluorouracil

SUMMARY:
RATIONALE: UCN-01 may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining UCN-01 with chemotherapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining UCN-01 with fluorouracil in treating patients who have metastatic pancreatic cancer that has not responded to treatment with gemcitabine.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate, time to progression, and overall survival of patients with gemcitabine-refractory metastatic pancreatic cancer treated with UCN-01 and fluorouracil.
* Determine the toxicity of this regimen in these patients.

OUTLINE: Patients receive fluorouracil IV over 24 hours on days 1, 8, 15, and 22. Patients also receive UCN-01 IV continuously over 72 hours (course 1 only) beginning on day 2. In subsequent courses, UCN-01 is infused over 36 hours. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study within 3-13 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas

  * Progressive disease after gemcitabine-based chemotherapy for metastatic disease
* At least 1 unidimensionally measurable metastatic lesion

  * At least 20 mm by conventional techniques OR
  * At least 10 mm by spiral CT scan
  * Primary disease site is not considered a measurable lesion
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1 OR
* Karnofsky 70-100%

Life expectancy

* More than 8 weeks

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin normal
* AST/ALT no greater than 2.5 times upper limit of normal

Renal

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac tachyarrhythmia

Pulmonary

* No symptomatic chronic obstructive pulmonary disease
* No pulmonary embolism within the past 6 months

Other

* No prior allergic reactions to compounds of similar chemical or biological composition to UCN-01 or other agents used in this study
* No diabetes mellitus uncontrolled by insulin or oral hypoglycemic agents
* No uncontrolled concurrent illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception before, during, and for 3 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy

Chemotherapy

* See Disease Characteristics
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No more than 1 prior chemotherapy regimen for metastatic or recurrent disease
* No prior fluorouracil in the adjuvant or inoperable, locally advanced setting (except as a radiosensitizer)
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* More than 4 weeks since prior radiotherapy and recovered
* No prior mediastinal irradiation
* No concurrent radiotherapy

Surgery

* Not specified

Other

* No prior UCN-01 or other cyclin-dependent kinase inhibitors
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational or commercial anticancer agents or therapies
* No concurrent anticonvulsant medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-07; Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary K. Schwartz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States